CLINICAL TRIAL: NCT03067415
Title: A Multi Center, Randomized, Double-blind, Parallel Design, Exploratory Trial to Evaluate the Efficacy and Safety of D565H Twice Daily Versus D565 Once Daily in Primary Open Angle Glaucoma or Ocular Hypertension Patients.
Brief Title: Exploratory Trial to Evaluate the Efficacy and Safety of D565H Twice Daily Versus D565 Once Daily
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 171GLC16020
Record Dates: First submitted 2017-02-24; First posted 2017-03-01 (Actual); Last update posted 2017-07-21 (Actual); Status verified 2017-02

CONDITIONS: Glaucoma, Primary Open Angle; Ocular Hypertension
Keywords: Glaucoma, Primary Open Angle; Ocular hypertension; CKD-351
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension

STUDY DESIGN:
Intervention Model Description: Assignment
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- D565H(Latanoprost 25㎍/㎖) (Experimental): D565H(Latanoprost 25㎍/㎖)
  Interventions: Drug: D565H(Latanoprost 25㎍/㎖); Drug: D565(Latanoprost 50㎍/㎖)
- D565(Latanoprost 50㎍/㎖) (Active Comparator): D565(Latanoprost 50㎍/㎖)
  Interventions: Drug: D565H(Latanoprost 25㎍/㎖); Drug: D565(Latanoprost 50㎍/㎖)

INTERVENTIONS:
Drug: D565H(Latanoprost 25㎍/㎖) — D565H twice daily
  Other Names: Arm A
Drug: D565(Latanoprost 50㎍/㎖) — D565 once daily
  Other Names: Arm B

SUMMARY:
Exploratory trial to evaluate the efficacy and safety of D565H twice daily versus D565 once daily.

DETAILED DESCRIPTION:
A Multi center, Randomized, Double-blind, Parallel design, Exploratory trial to evaluate the efficacy and safety of D565H twice daily versus D565 once daily in primary open angle glaucoma or ocular hypertension patients.

ELIGIBILITY:
Inclusion Criteria:

1. More than the age of 19 years old
2. Subjects who has primary Open-Angle Glaucoma or Ocular Hypertension
3. Subjects who sign on an informed consent form willingly

Exclusion Criteria:

1. Subjects with IOP(Intraocular Pressure) measured at Visit 1 and Visit 2(AM 09:00) above 35 mmHg at more than one eye
2. Subjects with a maximum corrected visual acuity of less or than 0.3 in the selected evaluation eye at visit 2
3. Subjects who were diagnosed as below with monocular or both eye

   * Acute or Chronic Closed-Angle Glaucoma
   * Secondary Glaucoma
   * Pseudoexfoliation Glaucoma
   * Neovascular Glaucoma
   * aphakia
   * phacocyst capsular torn intraocular lens
4. Subjects with significant eye symptoms/signs(Abscesses, diplopia) or severe visual field impairment(Mean Deviation -25dB or more)
5. Subjects with severe dry eye syndrome or progressive retinal disease(Retinal degeneration, Diabetic retinopathy, Retinal detachment, Macular edema)
6. Subjects with inflammatory/infectious eye disease and active eye disease within the last 3 months
7. Subjects who have medical history following

   * Glaucoma surgery
   * Subjects with significant history of ocular trauma during the last 6 months, or who underwent surgical ophthalmic surgery
   * Subjects who received topical or systemic steroids within the last 6 months
8. Subjects who wore need to wear contact lenses during the study
9. Subjects who have drug interaction with the investigational product, have a significant effect on the intraocular pressure, or who may have an effect on the clinical trial results
10. Subjects with known hypersensitivity to investigational product
11. Women who are nursing, pregnant or planning pregnancy during the study
12. Subjects with bronchial asthma or history
13. Subjects who have received any other investigational product within 1 month prior to the first dosing
14. Impossible subjects who participate in clinical trial by investigator's decision

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Estimated)
Dates: Start 2017-03-30 (Actual); Primary Completion 2017-09-10 (Estimated); Study Completion 2017-09-30 (Estimated)

PRIMARY OUTCOMES:
Change in mean intraocular pressure at 4 weeks compared to baseline | Baseline, 4 weeks
  Mean baseline intraocular pressure change Mean intraocular pressure change after 4 weeks

SECONDARY OUTCOMES:
Change in mean intraocular pressure at 2 weeks compared to baseline | Baseline, 2 weeks
  Mean baseline intraocular pressure change Mean intraocular pressure change after 2 weeks
Changes in intraocular pressure by measurement time | 2 weeks, 4 weeks
  IOP variation by measurement time

OTHER OUTCOMES:
Safety assessed by the incidence of adverse event, History, Medication | up to 4 weeks
  Adverse events, history, medications, signs of vitality, physical examination, etc.

CONTACTS AND LOCATIONS:
Overall Officials: KiHo Park, Principal Investigator — Seoul National University Hosipital
Locations (1):
- Seoul National University Hosipital, Seoul, Jongno, South Korea

IPD SHARING:
Plan to Share IPD: No